CLINICAL TRIAL: NCT00717301
Title: Accuracy of S-100B as Pre-Head CT Scan Screening Test After Mild Traumatic Brain Injury
Brief Title: S-100B as Pre-Head CT Scan Screening Test After Mild Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Academic Health Center Consortium (not Univ of Minnesota) (Unknown); New York State Department of Health (Other Government); Emergency Research Network of the Empire State (Unknown)
Responsible Party: Principal Investigator, Jeffrey Bazarian, Professor, University of Rochester
Other Study IDs: C806001
Record Dates: First submitted 2008-07-15; First posted 2008-07-17 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Traumatic Brain Injury
Keywords: TBI, traumatic brain injury, S100B, head CT scan
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Head Trauma: Patients presenting to any of the AHCC/ERNES Emergency Departments with head trauma.
- Control subjects: Patients presenting to the Univ of Rochester Medical Center/Strong Memorial Hospital Outpatient Laboratory for routine blood draw.

SUMMARY:
The purpose of the study is to determine if a specific blood protein, S-100B, can help predict who will have a traumatic abnormality on head CT scan after a concussion. We will compare the levels of this protein in the subject's blood to the initial head CT scan and to how the subject is feeling one month after injury. We hope that the information we collect in this trial will help us determine who needs a head CT scan after a concussion and who may be more likely to have trouble recovering from a concussion.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the ability of a serum S-100B to predict traumatic abnormalities on brain CT scan after mild traumatic brain injury (mild TBI). The secondary objective is to determine the relationship between initial S-100B levels and cognitive outcome at one month.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with head trauma to any of the AHCC/ERNES EDs, meeting the following criteria will be eligible to participate:

  * Presence of mild TBI per study definition
  * Arrival at the ED within 4 hours of injury
  * ED workup includes a Head CT

(Controls are eligible if they present to the Outpatient Lab for routine bloodwork during enrollment hours)

Exclusion Criteria:

* Time of injury not able to be determined
* Head CT not done as part of clinical emergency care
* Incarcerated
* Non-English or Spanish speakers
* Absence of parent/guardian for minor subjects
* Subject and/or parent/guardian do not have capacity to consent
* Head injury due to birth trauma, anoxia, inflammatory, toxic, infectious or metabolic encephalopathies that are not complications of head trauma
* Ischemic or hemorrhagic stroke without associated trauma

(Controls are excluded if they have any of the following:History of brain tumor, melanoma and/or Alzheimer's disease; History of concussion, bone fracture or stroke (CVA or TIA) in the past month; History of surgery in the past month; Inability to obtain consent from subject and/or parent due to lack of capacity or absence of parent/guardian of minor; Inability to speak or read English; Incarceration)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting to Emergency Departments that are a part of the AHCC (Academic Health Center Consortium) and/or ERNES (Emergency Research Network of the Empire State) networks.
Sampling Method: Non-Probability Sample
Enrollment: 1252 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Head CT scan | At time of injury in ED

SECONDARY OUTCOMES:
Post concussive symptoms | One month after injury

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Bazarian, MD, MPH, Principal Investigator — University of Rochester
Locations (6):
- United States (6):
  - Albany Medical College, Albany, New York
  - Erie County Medical Center, Buffalo, New York
  - Bassett Healthcare, Cooperstown, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical Center at Syracuse, Syracuse, New York
  - Guthrie, Sayre, Pennsylvania